CLINICAL TRIAL: NCT04158011
Title: CARs for CNS-Leukemia Relapse: A Retrospective International Study
Brief Title: A Retrospective Study of Patients With Leukemia Relapse in the CNS Treated With CAR T Cells
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Elad Jacoby, MD, Head, Pediatric Cancer Immunotherapy, Sheba Medical Center
Other Study IDs: SMC 6257-19
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: CAR T cells; CNS leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CNS ALL at lymphodepletion: Patients with active CNS leukemia at the time of lymphodepletion
- CNS ALL at inclusion: Patients who were referred to CAR T-cells with CNS disease, which was cleared by the time of lymphodepletion

SUMMARY:
CAR T cells targeting CD19 have been approved for patients with relapsed or refractory ALL, failing two or more prior protocols. Several institutional-based studies with other CAR T cells targeting CD19 have demonstrated outstanding response rates in patients with refractory disease, and the ability of CAR T cells to clear CNS leukemia. Nevertheless, these cases are sparse and have never been reported collectively.

Here, we aim to retrospectively assess toxicity and long term outcome of patients treated with CAR T cells for CNS relapse of ALL.

ELIGIBILITY:
Inclusion Criteria:

* Prior diagnosis of B-cell acute lymphoblastic leukemia involving the central nervous system
* Treatment with CAR T cells (either on a clinical trial or commercial use) due to this indication

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective review of patients with CNS - involvement of B-cell ALL, treated with CAR T cells targeting CD19 of either an institutional-based clinical trial, a pharma-based clinical trial or commercial product.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 6 months
  Duration between CAR T-cell infusion and death or last follow-up, according to Kaplan-Meier analysis

SECONDARY OUTCOMES:
Incidence of CAR-related CRS or ICANS per ASCTC guidelines | 2 months
  Number of patients and average grade of cytokine-release syndrome and immune-effector cell associated neurotoxicity syndrome within 2 months after CAR treatment, according to ASCTC guidelines (Lee et al, BBMT 2019)
Leukemia-free survival | 6 months
  Duration between CAR T-cell infusion and leukemia relapse, according to Kaplan-Meier analysis
CNS-leukemia free survival | 6 months
  Duration between CAR T-cell infusion and CNS leukemia relapse, according to Kaplan-Meier analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel